CLINICAL TRIAL: NCT03024177
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study of Vapendavir Treatment of Hematopoietic Stem Cell Transplant Subjects With Symptomatic Rhinovirus Infection
Brief Title: A Study of Vapendavir Treatment of Hematopoietic Stem Cell Transplant Subjects With Symptomatic Rhinovirus Infection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is withdrawn due to company decision
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BTA798-204
Record Dates: First submitted 2017-01-12; First posted 2017-01-18 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Rhinovirus; Upper Respiratory Tract Infection
Keywords: Human rhinovirus; HRV; Hematopoietic Stem Cell Transplant; HSCT; Antiviral; vapendavir; Allogeneic; Autologous
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vapendavir 528 mg (Experimental)
  Interventions: Drug: Vapendavir
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Vapendavir — Vapendavir Tablets, 264 mg
  Other Names: BTA798
  Arms: Vapendavir 528 mg
Drug: Placebo Oral Tablet — Vapendavir 264 mg matching tablets
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study of vapendavir treatment of laboratory-confirmed and symptomatic HRV infection of the upper respiratory tract in allogeneic and autologous stem cell transplant subjects. The aim of this study is to evaluate the effect of vapendavir on laboratory-confirmed HRV upper-respiratory tract infection in HSCT patients, as measured by viral load changes, worsening of upper respiratory tract infection (URTI) to lower respiratory tract infection (LRTI), duration of clinical symptoms, the occurrence of supplemental oxygen use, duration of viral shedding, hospital admission and duration of hospitalization, incidence of secondary bacterial infection, and mortality rates. Additionally, the safety and tolerability of vapendavir, and the vapendavir plasma levels achieved in the HSCT population, and the profile of viral resistance development will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Allogeneic or autologous HSC transplant within last 6 months using any conditioning regimen, or HSC transplant subjects with current chronic graft vs host disease requiring systemic treatment at any time point post-transplant;
2. Documented HRV in the upper respiratory tract (e.g., nasal swab, nasopharyngeal swab, nasal wash) as determined by local testing;
3. Subject presents to clinic reporting symptoms of a cold with the presence of at least 2 symptoms associated with HRV infection and with an onset such that they can be randomized and dosed preferably within 72 hours but up to a 5 day window (120 hours) interval from symptom onset to study treatment initiation;
4. Capable of giving written informed consent that includes compliance with the requirements and restrictions listed in the consent form. Informed consent and subject assent for subjects below the legal age of consent will be documented by means of a written, signed, and dated ICF and assent document. For subjects below the legal age of consent, the parent/legal guardian will provide informed consent and subjects below the legal age of consent will provide assent to participate in the study, in compliance with local regulations;
5. Subject is able to understand and comply with the protocol requirements;
6. Ability to maintain adequate oral intake of medication;
7. Female subjects who are not postmenopausal for at least 2 years or surgically sterile with complete hysterectomy or bilateral oophorectomy and male subjects, who are not surgically sterile via vasectomy, must agree to use a double barrier method of birth control, such as, a condom plus spermicidal agent (foam/gel/film/cream/suppository) from the time of randomization until 30 days after completion of study drug dosing. Male subjects cannot donate sperm during the study starting at day 1 and for 90 days after completion of study drug dosing;
8. Female subjects must not be breastfeeding or pregnant.

Exclusion Criteria:

1. Positive test result within 5 days prior to Study Day 1 inclusive for any of the following viral respiratory pathogen that are not HRV: respiratory syncytial virus, influenza, parainfluenza, adenovirus, or human metapneumovirus;
2. Clinically significant bacterial, fungal, or viral lower respiratory tract infection within 2 weeks prior to Study Day 1 (subject cannot have lower respiratory tract infection at Study Day 1) inclusive that has not been adequately treated, as determined by the investigator;
3. Clinically significant systemic bacteremia or fungemia within 7 days prior to Study Day 1 that has not been adequately treated, as determined by the investigator and the Medical Monitor;
4. Subjects receiving high dose systemic steroids defined as >2mg/kg per day or prednisone or prednisone equivalent currently or within the 7 days prior to Study Day 1;
5. Subjects with diagnosis of a lower respiratory infection at Study Day 1, subjects with O2 saturation of less than 92% in the absence of supplemental oxygen, or those requiring invasive mechanical ventilation or non-invasive mechanical ventilation with BIPAP or CPAP at the time of randomization, and/or a history or current evidence of chronic obstructive airways disease, emphysema, cystic fibrosis or current, uncontrolled or severe asthma;
6. Moderate to severe hepatic veno-occlusive disease (VOD), now known as moderate to severe sinusoidal obstructive syndrome (SOS), defined as meeting Baltimore Criteria for moderate or severe VOD disease;
7. At the time of randomization, currently in hospice, or at overt risk of death, in the judgment of the investigator. If relapsed with hematologic malignancy, subject may be enrolled if status not futile and subject expected at the time of randomization to survive to complete the study;
8. Subjects with absolute lymphocyte count of >2000 cells/mm3 within 5 days of randomization (Study Day 1);
9. Subjects with other known clinical significant laboratory abnormalities from local lab testing performed within 30 days prior to Study Day 1 will be considered for inclusion, if in the opinion of the investigator or Medical Monitor the abnormalities will not significantly jeopardize the safety of the subject or are related to the underlying study disease and/or transplant and the abnormalities will not impair the validity of the study;
10. Known history of estimated creatinine clearance < 50 mL/min (as calculated via the Cockcroft-Gault method);
11. Known history of HIV/AIDS. Known history of active HBV or HCV infection that has not resolved with treatment;
12. Current abuse of alcohol or any use of illicit drugs;
13. Received an investigational drug or investigational vaccine within 14 calendar days or 5 half-lives (whichever is longer) which does have US market approval for a related indication or different dosing regimen, or use of an investigational medical device within 14 calendar days prior to Study Day 1, or has received vapendavir at any previous time;
14. Subjects unable to tolerate bilateral nasopharyngeal sampling required for this study, as determined by the investigator.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Efficacy: Time-weighted average change from baseline to end of treatment visit in HRV viral load (HRV-RNA log10 copies/mL) | Study Day 1 to end of treatment (Study Day 14)
Safety: Proportion of treatment-emergent adverse events | Study Day 1 - 90
Safety: Proportion of treatment-related serious adverse events | Study Day 1 - 90
Safety: Incidence of treatment-emergent Grade 3 or greater clinical laboratory abnormalities | Study Day 1 - 90

CONTACTS AND LOCATIONS:
Overall Officials: Anna Novotney-Barry, Study Director — Aviragen Therapeutics, Inc.